CLINICAL TRIAL: NCT00572702
Title: Open, Randomized, Prospective, Comparative, Multicentric to Treat Prolapse of Vaginal Cuff After Hysterectomy With Amreich Procedure or Total Prolift Procedure
Brief Title: Randomized,Multicentric Study to Treat Prolapse After Hysterectomy With Amreich Procedure or Total Prolift Procedure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charles University, Czech Republic (Other)
Collaborators: Ministry of Health, Czech Republic (Other Government)
Responsible Party: prof. Michael Halaska, MD., PhD., Inner Grant Agency, Ministry of Health, Czech republic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NR/9309-3 IGA; NR/9309-3 IGA
Record Dates: First submitted 2007-12-12; First posted 2007-12-13 (Estimated); Last update posted 2009-08-03 (Estimated); Status verified 2009-07

CONDITIONS: Pelvic Organ Prolapse
Keywords: Biocompatible Materials; Female; Humans; Pelvic Floor; Polypropylenes; Prostheses and Implants; Surgical Mesh; Uterine Prolapse/*therapy
MeSH Terms: conditions — Pelvic Organ Prolapse

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Active Comparator): Patients with 3 compartment pelvic organ prolapse after hysterectomy, treated with Amreich-Richter procedure; it will be set randomly
  Interventions: Procedure: Vaginal fixation Amreich-Richter
- B (Active Comparator): Patients with 3 compartment pelvic organ prolapse after hysterectomy, treated with total Prolift procedure; it will be set randomly
  Interventions: Procedure: Prolift total

INTERVENTIONS:
Procedure: Vaginal fixation Amreich-Richter — Descending vaginal cuff will be treated with fixation of the cuff on sacrospinous ligament
  Arms: A
Procedure: Prolift total — Descending vaginal cuff will be treated with insertion of site-specific mesh into the vesico-vaginal and recto-vaginal space
  Other Names: Prolift total - polypropylen mesh
  Arms: B

SUMMARY:
Head to Head comparison of perioperative complications and secondary the impact of operation techniques with or without mesh on patients suffering from pelvic organ prolapse on quality of life.

DETAILED DESCRIPTION:
During the last decade a substantial progress in the detailed knowledge of morphology and function of different compartments of the female pelvic floor was achieved. The obtained informations were quickly implemented in the clinical practice especially in the application of special meshes and of novel techniques of their implantation. Their success rate was evaluated only in pilot companies supported studies. We do miss randomised studies not sponsored by company comparing different surgical techniques and their impact on the quality of life (QoL); the objective estimation of those consequences is for the longlasting effect of the surgery inevitable. The new methods bring also new complications which were not yet relevantly and objectively documented.

In the study we compare the techniques contemporary used - in the groups with or without mesh, in size relevant for the statistical evaluation

ELIGIBILITY:
Inclusion Criteria:

* female sex
* age 18 and more
* subscribed informed consent
* objective symptoms of prolapse-POP-Q 3 and more according to ICS standards
* compliance of the patient

Exclusion Criteria:

* patients with evidence of malignant lesion in small pelvis
* history of radiotherapy in small pelvis
* patients suffering from any form of PID within inclusion process
* pregnancy
* lactation
* total eversion of uterus and vagina
* serious internal disorders
* history of recto- or vesico-vaginal fistula
* history of rejection of any artificial material
* symptoms of primary genuine stress urinary incontinence
* patients who were not able to subscribe the informed consent
* patients, who couldn´t be reached for further follow-up

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2007-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
The objective evaluation o perioperative complications and comparison of patients with pelvic organ prolapse treated with Amreich-Richter procedure or Prolift implants. | 3 month

SECONDARY OUTCOMES:
Ultrasound, urodynamics, clinical examinations, magnetic resonance imaging, validated QoL questionnaires | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Michael Halaska, MD,PhD, Principal Investigator — Charles University, Prague, Czech Republic
Locations (5):
- Czechia (5):
  - Dpt. Obstetrics and gynecology, General Teaching Hospital, Prague
  - Institute for the care of mother and child, Prague
  - Dpt. of gynecology, Central military hospital, Prague
  - Dpt. Obstetrics and gynecology, Teaching hospital Bulovka, Prague
  - Dpt. of Obstetrics and gynecology, Bata hospital, Zlín